CLINICAL TRIAL: NCT06820151
Title: Characterising the Genomic and Phenotypic Changes That Define Injury and Repair in the Context of Early Carcinogenesis in the Human Oesophagus.
Brief Title: Exploring the Landscape of Injury and Repair in the Human Oesophagus
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 293952
Record Dates: First submitted 2025-01-29; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Perforations to the Oesophagus
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EVT sponges, tissue brushings and pinch biopsies from upper GI surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Group 1 will include patients who are having elective upper gastro-intestinal surgery where a leak is a recognised complication (but has not occurred).
  Interventions: Other: Sample collection
- Group 2: Group 2 will include patients who present acutely with an upper gastro-intestinal leak.
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Sample collection: EVT sponges, tissue brushings and pinch biopsies

SUMMARY:
The goal of this study limited to working with human tissue samples is to delineate the mechanisms defining appropriate oesophageal injury and repair and to use this information to understand how these rules are dysregulated and result in cancer formation in adult patients undergoing endoluminal vacuum therapy (EVT therapy) for the treatment of perforations to the oesophagus.

The main question[s] it aims to answer are:

* to gain a deeper understanding of the processes underlying tissue regeneration and repair in the oesophagus and upper gastro-intestinal tract following physical injury
* to identify the similarities in the processes of regeneration and early carcinogenesis

Participants will take part in the study during their usual EVT therapy schedule. Tissue brushings and pinch biopsies will also be taken.

DETAILED DESCRIPTION:
Tissue injury activates a number of cellular responses to initiate wound healing, resulting in the formation of new tissue within a short span of time and in a controlled fashion. In contrast, cancer results when a tissue mass forms in an unregulated process. Understanding the molecular mechanisms behind appropriate wound healing enables us to delineate how this process goes askew in the context of cancer. The goal is to delineate the mechanisms defining appropriate oesophageal injury and repair, and to use this information to understand how these rules are dysregulated and result in cancer formation.

In this study, the researchers wish to recruit adult patients undergoing endoluminal vacuum therapy (EVT therapy) for the treatment of perforations to the oesophagus in order to collect the discarded EVT sponge, biopsies from endoscopies, resected surgical specimens and additional blood samples. The researchers will request consent for access to archived tissue samples from any previous related surgery and some associated clinical metadata. The samples and associated clinical metadata will then be pseudonymised and sent to the Wellcome Sanger Institute.

Once samples are received at the Wellcome Sanger Institute, they will undergo a number of procedures including but not limited to genome sequencing, this will enable the researchers to gain a better understanding of the wound healing process, specifically how it can sometimes go wrong and lead to the development of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients 18 years old and over who are having elective upper gastro-intestinal surgery where a leak is a recognised complication (but has not occurred)
* Male and Female patients 18 years and over who present acutely with an upper gastro-intestinal leak.

Exclusion Criteria:

* patients who do not have a good understanding of the English Language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing endoluminal vacuum therapy (EVT) for the treatment of perforations to the oesophagus in order to collect the discarded EVT sponge, biopsies from endoscopies, resected surgical specimens and additional blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Genetic changes in regenerating oesophageal tissue | approximately 52 months
  To develop a detailed description of the genetic changes in regenerating oesophageal tissue in cancerous vs. non-cancerous oesophageal tissue
Characterising germline mutations | approximately 52 months
  blood samples will be used to characterise the 'germline mutations' or inherited mutations present in all of the participants cells. The samples will be processed to separate the white blood cells which will then undergo processes to look at individual genes, collections of genes, exomes, whole exomes and whole genome sequencing (WGS)
DNA sequencing | approximately 52 months
  DNA from microdissected and in vitro cultured tissues will be extracted and sequenced using state-of-the-art sequencing methods to look at individual genes, collections of genes, exomes, whole exomes and whole genomes.

CONTACTS AND LOCATIONS:
Overall Officials: AYESHA NOORANI, PhD MRCS, Principal Investigator — Genome Research Limited operating as The Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The Wellcome Sanger Institute never shares identifiable information about any of those who participate in its research and has strict measures in place to ensure that the privacy of research participants is protected.